CLINICAL TRIAL: NCT03603444
Title: Serum Calcium to Phosphorus (Ca/P) Ratio to Define Disorders of Ca-P Metabolism
Brief Title: Reliability of Serum Calcium to Phosphorus (Ca/P) Ratio as an Accurate and Inexpensive Tool to Define Disorders of Ca-P Metabolism
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Vincenzo Rochira, Professor, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 0032443/15
Record Dates: First submitted 2018-07-10; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Phosphorus and Calcium Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First study group: patients with PHPT: Patients aged between 18-90 years old with primary hyperparathyroidism who had been diagnosed in the Unit of Endocrinology of the University of Modena and Reggio Emilia.
  Exclusion criteria for both cases and controls will be: age younger than 18 or older than 90 years; severe renal and liver diseases (i.e. glomerular filtration rate (GFR) <30 ml/min); hyperparathyroidism secondary to Vitamin D deficiency; active metabolic bone disease (e.g. Paget's disease of the bone, osteomalacia, rickets, etc); any type of cancer; malnutrition; severe obesity (BMI > 40 kg/m2); a history of gastrointestinal malabsorption; sarcoidosis; hypercortisolism, diabetes insipidus, hyperthyroidism, pseudohypoparathyroidism; familial hypocalciuric hypercalcemia (FHH); treatment with steroids, active forms of vitamin D (calcitriol, ergocalciferol, etc), thiazides, phosphate binders, lithium, cinacalcet, bisphosphonates, and denosumab.
  Interventions: Other: No intervention are provided
- Second study group: patients with HypoP: Subjects with reduced serum P, but normal serum Ca, will be enrolled among HIV-infected patients on HAART treatment from the Modena cohort.
  Exclusion criteria for both cases and controls will be: age younger than 18 or older than 90 years; severe renal and liver diseases (i.e. glomerular filtration rate (GFR) <30 ml/min); hyperparathyroidism secondary to Vitamin D deficiency; active metabolic bone disease (e.g. Paget's disease of the bone, osteomalacia, rickets, etc); any type of cancer; malnutrition; severe obesity (BMI > 40 kg/m2); a history of gastrointestinal malabsorption; sarcoidosis; hypercortisolism, diabetes insipidus, hyperthyroidism, pseudohypoparathyroidism; familial hypocalciuric hypercalcemia (FHH); treatment with steroids, active forms of vitamin D (calcitriol, ergocalciferol, etc), thiazides, phosphate binders, lithium, cinacalcet, bisphosphonates, and denosumab.
  Interventions: Other: No intervention are provided
- Control group: Patients that underwent biochemical examination by primary care physician or by endocrinologist in order to assess their calcium-phosphorus metabolism state with normal results.
  Exclusion criteria for both cases and controls will be: age younger than 18 or older than 90 years; severe renal and liver diseases (i.e. glomerular filtration rate (GFR) <30 ml/min); hyperparathyroidism secondary to Vitamin D deficiency; active metabolic bone disease (e.g. Paget's disease of the bone, osteomalacia, rickets, etc); any type of cancer; malnutrition; severe obesity (BMI > 40 kg/m2); a history of gastrointestinal malabsorption; sarcoidosis; hypercortisolism, diabetes insipidus, hyperthyroidism, pseudohypoparathyroidism; familial hypocalciuric hypercalcemia (FHH); treatment with steroids, active forms of vitamin D (calcitriol, ergocalciferol, etc), thiazides, phosphate binders, lithium, cinacalcet, bisphosphonates, and denosumab.
  Interventions: Other: No intervention are provided

INTERVENTIONS:
Other: No intervention are provided

SUMMARY:
BACKGROUND: Primary hyperparathyroidism (PHPT) is the third most common endocrine disorder. The Ca/P ratio is an accurate tool to differentiate patients with PHPT (>3.5 if Ca and P are expressed in mg/dl) from healthy subjects. The reliability of this index is based on the fact that serum Ca and P are inversely related together. However, other disorders of the Ca-P metabolism, such as hypophosphoremia (HypoP) not related to PHPT, might also impair the Ca/P ratio.

OBJECTIVE: To validate the accuracy of Ca/P ratio in the diagnosis of Ca-P metabolism disorders, including also patients with documented HypoP not related to PHPT.

METHODS: A single-center, retrospective, case-control study will be carried out.

Biochemical measurements will include parathormone (PTH), vitamin D, serum Ca and P, serum albumin and creatinine.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of primary hyperparathyroidism
* HIV-infected patients with reduced phosphorus but normal calcium
* subjects with normal Calcium-Phosphorus metabolism

Exclusion criteria for both cases and controls will be:

* age younger than 18 or older than 90 years
* severe renal and liver diseases (i.e. glomerular filtration rate (GFR) <30 ml/min)
* hyperparathyroidism secondary to Vitamin D deficiency
* active metabolic bone disease (e.g. Paget's disease of the bone, osteomalacia, rickets, etc)
* any type of cancer
* malnutrition
* severe obesity (BMI > 40 kg/m2)
* a history of gastrointestinal malabsorption
* sarcoidosis
* hypercortisolism
* diabetes insipidus
* hyperthyroidism
* pseudohypoparathyroidism
* familial hypocalciuric hypercalcemia (FHH)
* treatment with steroids, active forms of vitamin D (calcitriol, ergocalciferol, etc), thiazides, phosphate binders, lithium, cinacalcet, bisphosphonates, and denosumab.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Serum Calcium to Phosphorus ratio will be compared among patients with different disorders of calcium-phosphorus metabolism (primary hyperparathyroidism and hypophosphoremia) and controls.
Sampling Method: Non-Probability Sample
Enrollment: 606 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Serum Calcium to Phosphorus ratio | Assessed only once at the diagnosis (from January 2005 to January 2018)
  Calculated formula (serum calcium to serum phosphorus ratio)

SECONDARY OUTCOMES:
Serum Calcium | Assessed only once at the diagnosis (from January 2005 to January 2018)
  From blood sample - Unit of measurement: mg/dl
Serum Phosphorus | Assessed only once at the diagnosis (from January 2005 to January 2018)
  From blood sample - Unit of measurement: mg/dl
Serum Parathormone | Assessed only once at the diagnosis (from January 2005 to January 2018)
  From blood sample - Unit of measurement: pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero - Universitaria di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No